CLINICAL TRIAL: NCT05146245
Title: Safety and Pharmacokinetics of Antipsychotics in Children 2: Studying TDM in an RCT
Acronym: SPACe2:STAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting de Merel (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Birgit Koch, Prof.Dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MEC-2021-0278; 2020-005450-18 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2021-12-06 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Risperidone; Therapeutic Drug Monitoring
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Drug Monitoring (Experimental): Physicians receive dosing advice based on measured blood levels of risperidone and 9-OH-risperidone.
  Interventions: Other: Therapeutic Drug Monitoring; Other: Risperidone plasma level
- Care As Usual (Active Comparator): Physician decides on possible dosing changes without receiving advice based on blood levels.
  Interventions: Other: Risperidone plasma level

INTERVENTIONS:
Other: Therapeutic Drug Monitoring — Physician receives dosing advice based on risperidone plasma level.
  Arms: Therapeutic Drug Monitoring
Other: Risperidone plasma level — Plasma levels of risperidone and 9-OH risperidone are measured in a Dried Blood Spot.

SUMMARY:
The aim of this study is to test whether therapeutic drug monitoring of risperidone in children with autism spectrum disorder and comorbid behavioral problems is able to reduce metabolic side effect burden, while retaining clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years
* Documented clinical diagnosis of autism spectrum disorder according to DSM IV or DSM V and comorbid behavioural problems
* To start treatment with risperidone

Exclusion Criteria:

* Diabetes type I or II
* Congenital or acquired syndrome associated with changes in appetite, body weight or lipid profile (e.g. Prader Willi)
* Treatment with antipsychotic medication within the last 6 months
* Known Long QT syndrome (LQTS)
* Pregnancy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
BMI z-score | 6 months
  Difference in body mass index z-scores 6 months after start of treatment.

SECONDARY OUTCOMES:
Effectivity (ABC) | 6 months
  Difference on the Irritability scale of the Aberrant Behavior Checklist (scores ranging from 0 to 45, a higher score means more symptoms) 6 months after start of treatment.
Effectivity (CGI) | 6 months
  Difference on the Clinical Global Impression scale (scores ranging from 1 to 7, a higher score means higher severity) 6 months after start of treatment.
Quality of Life (PedsQL) | 6 months
  Difference on Pediatric Quality of Life Inventory (scores ranging from 0 to 100, a higher score indicates a better quality of life) 6 months after start of treatment.
Metabolic side effects (glucose) | 6 months
  Difference in level of glucose 6 months after start of treatment.
Metabolic side effects (cholesterol) | 6 months
  Difference in levels of cholesterol and lipoproteins (LDL, HDL) 6 months after start of treatment.
Metabolic side effects (triglycerides) | 6 months
  Difference in level of triglycerides 6 months after start of treatment.
Endocrine side effects (prolactin) | 6 months
  Difference in level of prolactin 6 months after start of treatment.
Extrapyramidal symptoms (EPS) | 6 months
  Difference in extrapyramidal symptoms measured by Abnormal Involuntary Movement Scale 6 months after start of treatment.
Endocrine side effects (ghrelin) | 6 months
  Difference in level of ghrelin 6 months after start of treatment.
Endocrine side effects (leptin) | 6 months
  Difference in level of leptin 6 months after start of treatment.
Side effects (blood pressure) | 6 months
  Difference in diastolic and systolic blood pressure 6 months after start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hermans RA, Ringeling LT, Liang K, Kloosterboer SM, de Winter BCM, Hillegers MHJ, Koch BCP, Dierckx B. The effect of therapeutic drug monitoring of risperidone and aripiprazole on weight gain in children and adolescents: the SPACe 2: STAR (trial) protocol of an international multicentre randomised controlled trial. BMC Psychiatry. 2022 Dec 20;22(1):814. doi: 10.1186/s12888-022-04445-6. PMID 36539734